CLINICAL TRIAL: NCT03705416
Title: Reflux in the Obese Undergoing Surgery or Endoscopy (ROSE) Previously: Gastroesophageal Reflux Disease (GERD) in Bariatric Patients
Brief Title: Long Term Outcomes of Bariatric Patients Treated With Surgery or Endoscopy
Acronym: ROSE
Status: Active, not recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00186052; The ROSE study (Other: Johns Hopkins University)
Record Dates: First submitted 2018-09-21; First posted 2018-10-15 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: GERD; Obesity
Keywords: GERD; Bariatric surgery; Endoscopic sleeve gastroplasty; Sleeve gastrectomy; Roux-en-Y gastric bypass
MeSH Terms: conditions — Gastroesophageal Reflux; Obesity | interventions — Endoscopy; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endoscopic sleeve gastroplasty: All obese patients who will be undergoing an endoscopic sleeve gastroplasty (ESG). As part of the standard of care this patients will have a preoperative gastroscopy with wireless pH monitoring. Then after the endoscopic sleeve gastroplasty patients will be followed up regarding GERD symptoms for 5 years. As part of the standard of care a follow up endoscopy will be done at year 1 and wireless pH monitoring will be performed
  Interventions: Procedure: Endoscopy
- Surgery (VSG or RYGBP): All obese patients who will be undergoing either a vertical sleeve gastrectomy or a Roux-en-Y gastric bypass. As part of the standard of care this patients will have a preoperative gastroscopy with wireless pH monitoring. Then after the surgical procedure patients will be followed up regarding GERD symptoms for 5 years. As part of the standard of care a follow up endoscopy will be done at year 1 and wireless pH monitoring will be performed
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Endoscopy — endoscopic suturing of stomach
  Other Names: Endoscopic sleeve gastroplasty or ESG
  Groups: Endoscopic sleeve gastroplasty
Procedure: Surgery — Vertical sleeve gastrectomy (VSG) surgical reduction of stomach, or (RYGBP) , or gastric bypass procedure
  Other Names: Surgical reduction or bypass
  Groups: Surgery (VSG or RYGBP)

SUMMARY:
GERD is common in the obese population. Bariatric procedures are the mainstay of therapy for these patients. Bariatric procedures can be surgical (Roux-en-Y gastric bypass and Vertical sleeve gastrectomy) or endoscopic (endoscopic sleeve gastroplasty). The rate of GERD after either treatment is unknown as is the rate of silent reflux. The study primary objective is to assess the incidence rate of GERD in bariatric patients that undergo either therapy.

DETAILED DESCRIPTION:
GERD is a prevalent condition worldwide, estimated to be around 20-30 % in North America. Obesity is rapidly increasing with an estimated prevalence of 66% in the adult population in the United States. GERD symptoms are common in the obese population with data showing weekly GERD symptoms in 34.6% and erosive esophagitis 26.9% in people with BMI > 30 Kg/m2.

Presently, bariatric procedures are the only sustainable method to address morbid obesity and its resulting comorbidities. There are endoscopic and surgical bariatric procedures. The natural history of GERD symptoms in this population after undergoing a bariatric treatment is scarce or conflicting. Moreover, silent or asymptomatic GERD prevalence has not been well established preoperatively. Evaluation and documentation of GERD may potentially change the planned bariatric procedure and avoid unnecessary additional surgeries or procedures to address symptomatic post-operative GERD.

The investigators hypothesized that GERD is more prevalent in patients undergoing surgical bariatric procedures, specifically laparoscopic vertical sleeve gastrectomy (VSG). This multi-center, prospective, cohort study can potentially clarify current debatable data, based mostly on retrospective studies, and can help clinicians to select the most appropriate bariatric treatment for the patients. Most importantly, by selecting the best approach based on preoperative GERD studies it could prevent long term complications of GERD and further unnecessary procedures for the bariatric patient.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 30 Kg/m2
* Patients scheduled to undergo a bariatric weight loss procedure (endoscopic or surgical)
* Patients older than 18 years and younger than 75 years of age at time of consent
* Patients able to provide written informed consent on the Institutional review board (IRB) approved informed consent form
* Patients willing and able to comply with study requirements for follow-up

Exclusion Criteria:

* Any patient with BMI < 30 Kg/m2
* Patients treated with intragastric balloons.
* Pre-existing esophageal stenosis/stricture preventing advancement of an endoscope during screening/baseline Esophagogastroduodenoscopy (EGD)
* Esophageal, gastric or duodenal malignancy
* Severe medical comorbidities precluding endoscopy, or limiting life expectancy to less than 2 years in the judgment of the endoscopist
* Uncontrolled coagulopathy or inability to be off anticoagulation or anti-platelet medication (ASA, Plavix) for 1 week prior to and 2 weeks after each endoscopy
* Active fungal esophagitis
* Known portal hypertension, visible esophageal or gastric varices, or history of esophageal varices
* General poor health, multiple co-morbidities placing the patient at risk, or otherwise unsuitable for trial participation
* Pregnant or planning to become pregnant during period of study participation
* Patient refuses or is unable to provide written informed consent
* Prior bariatric treatment procedure
* Prior surgical or endoscopic anti-reflux procedure

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Obese patients with BMI 30 scheduled to undergo a bariatric interventions (endoscopic and surgical) at multiple academic medical centers in the United States offering both treatments.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-03-30 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with GERD based on symptoms, and abnormal acid exposure time and/or reflux esophagitis | 1 year
  GERD symptoms, esophageal acid exposure time and/or esophagitis

SECONDARY OUTCOMES:
Difference in BMI after the bariatric procedure | 5 years
  change in weight in Kg and height in m (BMI=Kg/m) before and after treatment
Reflux esophagitis | 5 years
  Incidence of GERD-related complications
GERD severity based on standardized Reflux Disease Questionnaire (RDQ) | 3,6,12,24,26,48, and 60 months post procedure
  GERD severity based on standardized Reflux Disease Questionnaire (RDQ) questionnaire (score 12-72; the greater the score, the greater the severity)
GERD severity as assessed by GERD-Health related quality of life (HRQL) score | 3,6,12,24,26,48, and 60 months post procedure
  GERD-Health related quality of life (HRQL) score (score 0-53; the greater the score,the worse the quality of life) will be used for this assessment
Percentage of participants on daily or twice daily PPI for GERD symptoms control, regardless of pH-monitoring results | 5 years
  Proportion of patients being treated with medication (PPI)
Percent of patients with abnormal esophageal acid exposure time > 6% defined by Bravo pH monitoring (96 hours) | 1 year
  Abnormal esophageal acid exposure time (AET)
Percentage of excess body weight (EBW) loss and total body weight loss (TBWL) | 5 years
  Change in body weight after treatment with endoscopy and surgery (compare groups)
Prevalence and incidence of silent reflux | 1 year
  Proportion of patients with abnormal AET without symptoms after bariatric treatment procedure
Percentage of patients with GERD at baseline in whom the planned bariatric intervention was changed due to abnormal ph testing or presence of erosive esophagitis, Barrett's esophagus, reflux related esophageal stricture | 1 year
  Proportion of patients with change in treatment plan after diagnostic evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Marcia I Canto, MD, Principal Investigator — Johns Hopkins University
Locations (6):
- United States (6):
  - Johns Hopkins University, Baltimore, Maryland
  - Northwell Health, New Hyde Park, New York
  - Weill Cornell, New York, New York
  - Legacy Oregon Clinic, Portland, Oregon
  - Memorial Hermann Health System, Houston, Texas
  - Utah-Health: University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Research projects will be submitted to host (currently JHU) and accepted project will be granted access to read only de-identified database.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: available in 6 years
Access Criteria: Project submission to PI and or Heartburn Registry management team then if project accepted, security clearance and enrollment in REDCap and tutorial completions.

REFERENCES:
- [Background] Vakil N, van Zanten SV, Kahrilas P, Dent J, Jones R; Global Consensus Group. The Montreal definition and classification of gastroesophageal reflux disease: a global evidence-based consensus. Am J Gastroenterol. 2006 Aug;101(8):1900-20; quiz 1943. doi: 10.1111/j.1572-0241.2006.00630.x. PMID 16928254
- [Background] Tutuian R. Obesity and GERD: pathophysiology and effect of bariatric surgery. Curr Gastroenterol Rep. 2011 Jun;13(3):205-12. doi: 10.1007/s11894-011-0191-y. PMID 21424733
- [Background] Singh M, Lee J, Gupta N, Gaddam S, Smith BK, Wani SB, Sullivan DK, Rastogi A, Bansal A, Donnelly JE, Sharma P. Weight loss can lead to resolution of gastroesophageal reflux disease symptoms: a prospective intervention trial. Obesity (Silver Spring). 2013 Feb;21(2):284-90. doi: 10.1002/oby.20279. PMID 23532991
- [Background] Borbely Y, Schaffner E, Zimmermann L, Huguenin M, Plitzko G, Nett P, Kroll D. De novo gastroesophageal reflux disease after sleeve gastrectomy: role of preoperative silent reflux. Surg Endosc. 2019 Mar;33(3):789-793. doi: 10.1007/s00464-018-6344-4. Epub 2018 Jul 12. PMID 30003346
- [Background] El-Serag HB, Graham DY, Satia JA, Rabeneck L. Obesity is an independent risk factor for GERD symptoms and erosive esophagitis. Am J Gastroenterol. 2005 Jun;100(6):1243-50. doi: 10.1111/j.1572-0241.2005.41703.x. PMID 15929752
- [Background] Kurian M, Kroh M, Chand B, Mikami D, Reavis K, Khaitan L. SAGES review of endoscopic and minimally invasive bariatric interventions: a review of endoscopic and non-surgical bariatric interventions. Surg Endosc. 2018 Oct;32(10):4063-4067. doi: 10.1007/s00464-018-6238-5. Epub 2018 May 29. PMID 29845397
- [Background] Chung AY, Thompson R, Overby DW, Duke MC, Farrell TM. Sleeve Gastrectomy: Surgical Tips. J Laparoendosc Adv Surg Tech A. 2018 Aug;28(8):930-937. doi: 10.1089/lap.2018.0392. Epub 2018 Jul 13. PMID 30004814
- [Background] Schlottmann F, Buxhoeveden R. Laparoscopic Roux-en-Y Gastric Bypass: Surgical Technique and Tips for Success. J Laparoendosc Adv Surg Tech A. 2018 Aug;28(8):938-943. doi: 10.1089/lap.2018.0393. Epub 2018 Jul 16. PMID 30010475
- [Background] Rebecchi F, Allaix ME, Giaccone C, Ugliono E, Scozzari G, Morino M. Gastroesophageal reflux disease and laparoscopic sleeve gastrectomy: a physiopathologic evaluation. Ann Surg. 2014 Nov;260(5):909-14; discussion 914-5. doi: 10.1097/SLA.0000000000000967. PMID 25379861
- [Background] Burgerhart JS, Schotborgh CA, Schoon EJ, Smulders JF, van de Meeberg PC, Siersema PD, Smout AJ. Effect of sleeve gastrectomy on gastroesophageal reflux. Obes Surg. 2014 Sep;24(9):1436-41. doi: 10.1007/s11695-014-1222-1. PMID 24619293
- [Background] Oor JE, Roks DJ, Unlu C, Hazebroek EJ. Laparoscopic sleeve gastrectomy and gastroesophageal reflux disease: a systematic review and meta-analysis. Am J Surg. 2016 Jan;211(1):250-67. doi: 10.1016/j.amjsurg.2015.05.031. Epub 2015 Aug 14. PMID 26341463